CLINICAL TRIAL: NCT01978054
Title: Disseminating Evidence-Based Interventions to Control Cancer
Brief Title: Disseminating Public Health Evidence to Support State Health Department Prevention of Cancer and Other Chronic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201111105; 5R01CA160327 (NIH)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Information Dissemination; Evidence-Based Public Health
Keywords: Information Dissemination; Information Sharing; Innovation Diffusion; Public Health Practice; Evidence-Based Public Health; Chronic Disease Prevention; Cancer Prevention and Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dissemination (Experimental): Dissemination of public health knowledge: Participating states will help develop and choose 3-5 dissemination strategies they prefer for their state health department chronic disease units to receive. Dissemination strategies may include multi-day in-person training workshops, electronic information exchange modalities, and information on ways to enhance organizational climates favorable to evidence-based chronic disease prevention.
  Interventions: Other: Dissemination of public health knowledge
- Comparison (No Intervention): Comparison state health department chronic disease units will be provided links to preexisting sources of public health evidence-based information such as the Community Guide, Cancer Control P.L.A.N.E.T. (Plan, Link, Act, Network, with Evidence-based Tools), and NCI Research to Reality.

INTERVENTIONS:
Other: Dissemination of public health knowledge — State health department chronic disease units will be involved with developing and choosing dissemination activities to spread public health knowledge and information on population-based public health strategies that have been shown to reduce risk factors for cancer and other chronic diseases. Example of activities include: multi-day in-person training workshops and electronic information exchange modalities.
  Arms: Dissemination

SUMMARY:
The purpose of this study is to identify and evaluate dissemination strategies to promote the uptake of evidence-based cancer and other chronic disease prevention among state-level public health practitioners. Dissemination strategies such as multi-day in-person training workshops and electronic information exchange modalities are hypothesized to associate with improved access and use of public health evidence and organizational supports for program and policy decision making based on evidence-based public health.

DETAILED DESCRIPTION:
Evidence-based public health approaches to prevent cancer and other chronic diseases have been identified in recent decades and have the potential for high impact. Yet barriers to implement prevention approaches persist as a result of multiple factors including lack of organizational support, limited resources, competing priorities, and limited skill among the public health workforce. The purpose of this study was to learn how best to promote the adoption of evidence based public health practice related to chronic disease prevention. This cluster randomized trial aimed to evaluate the dissemination of public health knowledge about evidence-based prevention of cancer and other chronic diseases and test receptivity and usefulness of dissemination strategies directed toward state health department chronic disease practitioners to enhance capacity and organizational support for evidence-based chronic disease prevention. Twelve state health department chronic disease units were randomly selected and assigned to intervention or control. State health department staff and the university-based study team jointly identified, refined, and selected dissemination strategies. Intervention strategies included multi-day in-person training workshops, remote telephone follow-up and technical assistance, supplemental brief remote trainings, and health department work unit procedural changes to support and strengthen evidence-based decision making. Evaluation methods included pre-post surveys and structured qualitative phone interviews.

ELIGIBILITY:
Inclusion Criteria:

* State Health Department chronic disease units (cluster) in the United States and corresponding public health workforce (individuals within cluster)

Exclusion Criteria:

* State health department has received extensive technical assistance and training comparable to our intervention (dissemination activities)
* Origin state has no logical matching pair matched state based on state population size
* Origin state has the lowest excess burden of cancer and other chronic risk and disease
* Origin state health department has lowest or highest capacity for EBDM as determined from previous research

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1703 (Actual)
Dates: Start 2013-09; Primary Completion 2016-11 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Organizational supports for evidence-based decision making (EBDM) | 18-24 months post baseline
  Self-report Likert scale items in 4 factors: access to evidence and skilled staff, program evaluation, supervisory expectations and incentives for EBDM, and participatory decision-making

SECONDARY OUTCOMES:
EBDM competencies | 18-24 months post baseline
  Self-report Likert scale items measure perceived importance and availability of specific public health practitioner skill sets for EBDM
Use of research evidence for job tasks | 18-24 months post baseline
  Self-report frequency items for 6 job tasks, summary variable creating by calculating the mean frequency across the tasks

CONTACTS AND LOCATIONS:
Overall Officials: Ross C Brownson, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Prevention Research Center in St. Louis, Brown School, Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Survey participants were not asked for permission to share their unidentified data when data were first collected in 2014.

REFERENCES:
- [Derived] Jacob RR, Baker EA, Allen P, Dodson EA, Duggan K, Fields R, Sequeira S, Brownson RC. Training needs and supports for evidence-based decision making among the public health workforce in the United States. BMC Health Serv Res. 2014 Nov 14;14:564. doi: 10.1186/s12913-014-0564-7. PMID 25398652
- [Derived] Allen P, Sequeira S, Jacob RR, Hino AA, Stamatakis KA, Harris JK, Elliott L, Kerner JF, Jones E, Dobbins M, Baker EA, Brownson RC. Promoting state health department evidence-based cancer and chronic disease prevention: a multi-phase dissemination study with a cluster randomized trial component. Implement Sci. 2013 Dec 13;8:141. doi: 10.1186/1748-5908-8-141. PMID 24330729
- See also: Click here for more information about this study: Strategies in Disseminating Evidence — http://prcstl.wustl.edu
- See also: Study protocol entitled "Promoting state health department evidence-based cancer and chronic disease prevention: a multi-phase dissemination study with a cluster randomized trial component" — http://www.implementationscience.com/content/pdf/1748-5908-8-141.pdf
- See also: Intervention effects primary and secondary outcomes from pre-post survey data — https://www.cdc.gov/pcd/issues/2017/17_0326.htm
- See also: Organizational support associations with research evidence use in state public health agency chronic disease prevention units — https://journals.lww.com/jphmp/Abstract/publishahead/Organizational_Supports_for_Research_Evidence_Use.99481.aspx
- See also: Manager perspectives on organizational supports for evidence-based public health from interviews — https://link.springer.com/article/10.1007/s10900-018-0494-0